CLINICAL TRIAL: NCT01505920
Title: Lidocaine Spray Compared With Submucosal Injection in Reducing Pain During Loop Electrosurgical Excision Procedure: a Randomized Controlled Trial
Brief Title: Lidocaine Spray Compared With Submucosal Injection During LEEP: a Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, M.D., Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OBG-11-08-15A-12
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Uterine Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine spray (Experimental): 10% lidocaine spray 40 mg applied directly to the cervix, 3 minutes before starting cervical excision
  Interventions: Procedure: Lidocaine spray
- Lidocaine submucosal injection (Active Comparator): 2% lidocaine with 1:100,000 adrenaline 2 ml injected submucosally to the four quadrant of the cervix, 3 minutes before starting cervical excision
  Interventions: Procedure: Lidocaine submucosal injection

INTERVENTIONS:
Procedure: Lidocaine spray — 10% lidocaine spray 40 mg applied directly to the cervix, 3 minutes before starting cervical excision
  Arms: Lidocaine spray
Procedure: Lidocaine submucosal injection — 2% lidocaine with 1:100,000 adrenaline 2 ml injected submucosally into the four quadrant of the cervix, 3 minutes before starting cervical excision
  Arms: Lidocaine submucosal injection

SUMMARY:
Loop Electrosurgical Excision Procedure (LEEP) is a widely used minor surgical procedure for diagnosis and treatment of cervical intraepithelial neoplasia. During the procedure, several methods have been proposed to reducing pain including submucosal block, paracervical block, and oral analgesics. Submucosal (underneath the lining of the cervix) injection of lidocaine appeared to be the most common methods used. However, from the investigators experience, there is significant pain associated with the injection itself.

Lidocaine spray is an effective measure for pain control during minor gastrointestinal and otolaryngological procedures. It is simple without pain related to application.

An objective of this study is to examine effectiveness of lidocaine spray versus lidocaine submucosal injection by comparing pain scores at various stages of the LEEP procedure.

ELIGIBILITY:
Inclusion Criteria:

* Any degrees of cervical dysplasia detected from cervical cytology or histology
* Need to have loop electrosurgical excision procedure (LEEP) for diagnosis and/or treatment

Exclusion Criteria:

* Allergy to lidocaine
* Pregnancy
* Previous history of cervical operation including conization, LEEP, laser therapy and cryotherapy
* Cardiac arrhythmia
* Neural disease with impaired sensation
* Lower urinary tract cancer
* Coagulation defect
* Drug dependence
* Lower genital tract infection
* Obvious invasive disease of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Visual analog pain scores immediately after the excision | Immediately after the excision

SECONDARY OUTCOMES:
Visual analog pain scores at the time of anesthetic application | At the time of anesthetic application
Visual analog pain scores at 30 minutes after the procedure | At 30 minutes after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, M.D., Principal Investigator — Chiang Mai University; Asama Vanichtantikul, M.D., Principal Investigator — Chiang Mai University
Locations (1):
- Department of OB-GYN, Faculty of Medicine, Chiang Mai University, Chiang Mai, Chiang Mai, Thailand

REFERENCES:
- [Derived] Vanichtantikul A, Charoenkwan K. Lidocaine spray compared with submucosal injection for reducing pain during loop electrosurgical excision procedure: a randomized controlled trial. Obstet Gynecol. 2013 Sep;122(3):553-7. doi: 10.1097/AOG.0b013e31829d888e. PMID 23921860